CLINICAL TRIAL: NCT01701843
Title: A Phase II Exploratory Study Evaluating the Efficacy of Topical Cromoglicate Solution Compared to Topical Solution Vehicle in the Treatment of Mastocytosis
Brief Title: Cromoglicate in Mastocytosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: prematurely terminated because of low recruitment
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0074-33
Record Dates: First submitted 2012-07-11; First posted 2012-10-05 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2013-03

CONDITIONS: Mastocytosis
MeSH Terms: conditions — Mastocytosis | interventions — Cromolyn Sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (left) / Cromoglicate (right) (Other): Placebo (on a lesion left bodyside), Cromoglicate (on a lesion on right bodyside)
  Interventions: Drug: Cromoglicate; Drug: Placebo
- Placebo (right) / Cromoglicate (left) (Other): Placebo (on a lesion right bodyside), Cromoglicate (on a lesion on left bodyside)
  Interventions: Drug: Cromoglicate; Drug: Placebo

INTERVENTIONS:
Drug: Cromoglicate — Twice daily topical treatment for 14 days
Drug: Placebo — Twice daily topical treatment for 14 days

SUMMARY:
The purpose of this exploratory study is to investigate the clinical efficacy of study drug (LP0074) in the treatment of Mastocytosis. The trial will be performed as a left/right comparison study in male/female subjects with mastocytosis, in a prospective, double-blinded, randomised, single centre setting.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent has been obtained
* Chronic stable symptomatic maculopapulous cutaneous mastocytosis or indolent systemic mastocytosis with skin involvement and a positive Darier's Sign
* Age between 18 and 70 years
* Either sex
* Any race or ethnicity
* Attending hospital outpatient clinic or the private practice of a dermatologist.

Exclusion Criteria:

* The presence of autoimmune and infectious disease including aggressive systemic mastocytosis
* Medical history or presence of epilepsy, significant neurological disorders, cerebrovascular attacks or ischemia
* Medical history or presence of myocardial infarction or cardiac arrhythmia which requires drug therapy, hyper/hypokalemia
* Evidence of severe renal dysfunction (creatinine > 1,5 times upper reference value)
* Evidence of significant hepatic disease (liver enzymes > 2 times upper reference value)
* Presence of active cancer which requires chemotherapy or radiation therapy
* Commitment to an institution in terms of § 40 Abs. 1 S. 3 Nr. 4 AMG
* Intake of antihistamines or leukotriene antagonists within 7 days prior to the beginning of the study
* Intake of oral corticosteroids within 14 days prior to randomisation
* Use of depot corticosteroids or chronic systemic corticosteroids within 21 days prior to randomisation
* Radiation therapy of target areas including UV therapy within 4 weeks prior to randomisation
* Confounding other dermatological diseases or conditions that can affect the symptoms of the target areas
* Known or suspected hypersensitivity to component(s) of investigational products.
* Current participation in any other interventional clinical trial.
* Subjects who have received treatment with any nonmarketed drug substance (i.e. an agent which has not yet been made available for clinical use following registration) within the last 4 weeks or 5 half-lives (whichever is longer) prior to randomisation
* Previously randomised in this clinical trial
* In the opinion of the investigator, the subject is unlikely to comply with the Clinical Study Protocol (e.g. alcoholism, drug dependency or psychotic state).
* Females who are pregnant, of child-bearing potential and wishing to become pregnant during the trial or are breast feeding.
* Females of child-bearing potential with positive pregnancy test at visit 1.
* Subjects (or their partner) not using an adequate method of contraception (according to national requirements, as applicable)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of mechanically induced changes of lesions | Baseline to week 2

SECONDARY OUTCOMES:
Evaluation of mechanically induced wheal and flare response | Baseline to week 2

CONTACTS AND LOCATIONS:
Overall Officials: Frank Siebenhaar, MD, Principal Investigator — Allergie-Centrum-Charité
Locations (1):
- Allergie-Centrum-Charité, Department of Dermatology and Allergy, Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No